CLINICAL TRIAL: NCT04642781
Title: Measurement of Eye Movements While Reading a German Text
Status: Completed | Type: Observational
Sponsor: University of Basel (Other)
Responsible Party: Principal Investigator, Anja Palmowski-Wolfe, Professor Dr. med., University of Basel
Other Study IDs: 2018-00283
Record Dates: First submitted 2020-11-18; First posted 2020-11-24 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Healthy Children

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthy children aged 8-13years (schoolgrade 2-5): Primary school children are asked to read a German text presented on a laptop screen
  Interventions: Diagnostic Test: reading of a text

INTERVENTIONS:
Diagnostic Test: reading of a text — Reading of 2 IRest Texts presented on a laptop in randomized order while eye movements are recorded with a tracking bar.

SUMMARY:
To establish normative value for reading parameters in healthy children of primary school age and in grades 2-5.

DETAILED DESCRIPTION:
Following initial assessment of feasibility, recruitment is expanded to children attending grades 2-5 recruited from 4 different primary schools in German speaking Switzerland. Two texts of The New International Reading Speed Test (IReST) of similar difficulty are presented on a laptop in randomized order. Children are asked to read the text aloud while eye movements are recorded with an eye tracking bar. The following parameters are analysed: reading speed (words/minute), number of saccades, number of fixations.

ELIGIBILITY:
Inclusion Criteria:

* 8-13 years
* child consent
* parental consent

Exclusion Criteria:

* unability to read

Ages: 8 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: children recruited from 4 primary schools in German speaking Switzerland
Sampling Method: Non-Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2018-03-30 (Actual); Primary Completion 2019-12-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Reading speed | 21 months
  words read per minute
number of saccades and fixations | 21 months
  how stable are the eyes while reading out loud

CONTACTS AND LOCATIONS:
Overall Officials: Anja M Palmowski-Wolfe, Prof, Principal Investigator — University Basel, University Eye Hospital Basel
Locations (1):
- University Basel, University Eye Hospital Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No
Sharing through publication

REFERENCES:
- [Result] Wertli J, Schotzau A, Trauzettel-Klosinski S, Palmowski-Wolfe A. Feasibility of Eye Movement Recordings with the SMI Tracking Bar in 10- to 11-Year-Old Children Performing a Reading Task. Klin Monbl Augenheilkd. 2020 Apr;237(4):510-516. doi: 10.1055/a-1101-9204. Epub 2020 Apr 24. PMID 32330981
- [Result] Wertli J, Schotzau A, Palmowski-Wolfe A. The Influence of Age on Eye Movements during Reading in Early Elementary School Children. Klin Monbl Augenheilkd. 2023 Apr;240(4):591-598. doi: 10.1055/a-2045-7271. Epub 2023 Apr 25. PMID 37164411